CLINICAL TRIAL: NCT04696510
Title: Biomarker Identification to Predict the Evolution of Migraine From an Episodic to a Chronic Condition
Brief Title: Physiopathology, Diagnosis and Therapy of Primary Cephalalgia and Adaptive Disorders
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IMAGO2020
Record Dates: First submitted 2020-12-21; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-11

CONDITIONS: Migraine
Keywords: Episodic migraine; Chronic migraine; Medication overuse; Nitroglycerin; fMRI
MeSH Terms: conditions — Migraine Disorders; Prescription Drug Overuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic migraineurs: This group includes patients with chronic migraine.
- Control group: This group includes healthy subjects.
- Episodic migraineurs: This group includes patients with episodic migraine

SUMMARY:
The main aim of the present pilot study is to prove the possibility to use the Nitroglycerin (NTG) model to describe the pathophysiology of headache using task-free advanced Magnetic Resonance Imaging (MRI) techniques, in order to depict the static changes of the ictal and inter-ictal phase of migraine attacks vs the pain free state in healthy subjects and to compare that with the spontaneous headache attack experienced by chronic migraineurs.

DETAILED DESCRIPTION:
Resting state functional magnetic resonance imaging (rs-fMRI) has depicted cyclical functional connectivity changes during the ictal and inter-ictal phase of the migraine attack. In this pilot study, Functional Connectivity (FC) changes during nitroglycerin (NTG) induced migraine attacks were assessed vs the pain-free condition in healthy subjects.

To this end, subjects with episodic migraine (EM) without aura were enrolled. NTG-triggered a spontaneous-like migraine attack in the subjects. They underwent 4 rs-fMRI scan repetitions during different phases of the attack (baseline, prodromal, full blown, recovery phase) with a 3 Tesla MR scanner. According to the pain field literature, several regions of interests were studied, in particular the thalamic areas and the salience network (SN) were selected as primary areas of interest for the analyses. Subjects' rs-fMRI data were first processed with a seed-based correlation analysis (SCA) to assess the static changes in FC between the thalamus and the rest of the brain during the experiment. The wavelet coherence approach (WCA) were also applied to test the changes in time-in-phase coherence between the thalamus and the salience network (SN).

Healthy subject were administered nitroglycerin as well and scanned at a pain free baseline and after 3 hours in order to compare the response.

The rebound headache that followed acute drug withdrawal were used as a surrogate paradigm of spontaneous attack. Patients with chronic migraine and medication overuse were hospitalized for a supervised withdrawal program at the Mondino Foundation; during the program if they experienced a rebound headache attack, they were scanned with a rs-fMRI acquisition.

The acquired imagines were analyzed with the same procedure regarding the evaluation of static and dynamic functional connectivity fluctuation.

ELIGIBILITY:
Episodic migraineurs

Inclusion Criteria:

* age between 18-60 years;
* diagnosis of episodic migraine without aura developed before the age of 50;
* no current prophylactic treatment for migraine prevention;
* chronic migraineurs with medication overuse according to the ICHDIII criteria

Exclusion Criteria:

* chronic or medication-overuse headache or cluster headache diagnosis;
* any chronic pain condition or disorders other than migraine;
* an alleged diagnosis of major psychiatric disorders such as depression, bipolar affective disorder and schizophrenia;
* a diagnosis of tension type headache with a frequency of more than 5 days per month;
* any cardiovascular diseases in which the NTG use could be contraindicated;
* blood pressure hypotension, closed angle glaucoma, anaemia;
* women in child bearing, breast feeding; continuous use of benzodiazepines;
* any neuroradiological pathological findings at a previous MRI scan of the head.

Chronic migraineurs

Inclusion Criteria:

* age between 18-60 years;
* diagnosis of migraine without aura developed before the age of 50 according to the ICHD III criteria;
* currently chronic migraineurs with medication overuse according to The International Classification of Headache Disorders 3rd edition (ICHDIII) criteria.

Exclusion Criteria:

* any chronic pain condition or disorders other than migraine;
* an alleged diagnosis of major psychiatric disorders such as depression, bipolar affective disorder and schizophrenia;
* a diagnosis of tension type headache with a frequency of more than 5 days per month;
* any cardiovascular diseases in which the NTG use could be contraindicated;
* blood pressure hypotension, closed angle glaucoma, anaemia; women in child bearing, breast feeding;
* continuous use of benzodiazepines;
* any neuroradiological pathological findings at a previous MRI scan of the head.

Healthy subjects

Inclusion Criteria:

* age between 18-60 years;
* overall good clinical condition, no neurological findings at the physical examination.

Exclusion criteria:

* history of episodic or chronic or medication-overuse headache or cluster headache diagnosis according to the International Chronic Headache Disease (ICHD) III criteria;
* any chronic pain condition or disorders other than migraine;
* an alleged diagnosis of major psychiatric disorders such as depression, bipolar affective disorder and schizophrenia;
* a diagnosis of tension type headache with a frequency of more than 5 days per month;
* any cardiovascular diseases in which the NTG use could be contraindicated;
* blood pressure hypotension, closed angle glaucoma, anaemia;
* women in child bearing, breast feeding;
* continuous use of benzodiazepines;
* any neuroradiological pathological findings at the baseline MRI scan of the head.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with episodic migraine without aura; patients with chronic migraine and medication overuse; healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Functional Connectivity (FC) changes | Up to 6 hours
  Functional connectivity pattern of changes profiling the different condition of the migraine experience. To depict the static and dynamics changes of brain activity during a migraine attack; ii) To validate the use of the NTG-induced attacks paradigm as a reliable instrument combined with an fMRI approach to compare the induced vs the spontaneous attack; iii) To describe possible differences in brain activity between attacks in chronic and episodic migraineurs.

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | Up to 6 hours
  To acquire sufficient MRI to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms. This can be achieved by combining clinical, psychological, biological, neurophysiological and MRI-derived features into a multimodal multi-parametric approach suitable for patient's classification. The ML and DL approaches could also be adopted to predict chronification, as well as the response to a withdrawal program for medication overuse headache.
Monthly migraine frequency (day/month) | Up to 6 hours
  To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.
Disease duration (years) | Up to 6 hours
  To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.
Nausea (number) | Up to 6 hours
  As a feature of the migraine attack.To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.
Vomiting (number) | Up to 6 hours
  As a feature of the migraine attack.To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.
Photophobia (number) | Up to 6 hours
  As a feature of the migraine attack.To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.
Phonophobia (number) | Up to 6 hours
  To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.
Aggravation by movement (number) | Up to 6 hours
  As a feature of the migraine attack. To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.
Throbbing pain (number) | Up to 6 hours
  As a feature of the migraine attack. To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.
Abortive medication (number of intake/month) | Up to 6 hours
  To acquire clinical data to identify feature patterns that can profile patient's condition using machine learning (ML) and deep learning (DL) algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, Prof, Principal Investigator — IRCCS Mondino Foundation, Pavia
Locations (1):
- Headache Science Center, Pavia, Italy

REFERENCES:
- [Background] Karsan N, Bose PR, O'Daly O, Zelaya FO, Goadsby PJ. Alterations in Functional Connectivity During Different Phases of the Triggered Migraine Attack. Headache. 2020 Jul;60(7):1244-1258. doi: 10.1111/head.13865. Epub 2020 Jun 22. PMID 32568433
- [Background] Thomsen LL, Kruuse C, Iversen HK, Olesen J. A nitric oxide donor (nitroglycerin) triggers genuine migraine attacks. Eur J Neurol. 1994 Sep;1(1):73-80. doi: 10.1111/j.1468-1331.1994.tb00053.x. PMID 24283432
- [Background] Schulte LH, May A. Functional Neuroimaging in Migraine: Chances and Challenges. Headache. 2016 Oct;56(9):1474-1481. doi: 10.1111/head.12944. Epub 2016 Sep 22. PMID 27654831
- [Background] Amin FM, Hougaard A, Magon S, Sprenger T, Wolfram F, Rostrup E, Ashina M. Altered thalamic connectivity during spontaneous attacks of migraine without aura: A resting-state fMRI study. Cephalalgia. 2018 Jun;38(7):1237-1244. doi: 10.1177/0333102417729113. Epub 2017 Aug 30. PMID 28853611
- [Background] Maniyar FH, Sprenger T, Monteith T, Schankin C, Goadsby PJ. Brain activations in the premonitory phase of nitroglycerin-triggered migraine attacks. Brain. 2014 Jan;137(Pt 1):232-41. doi: 10.1093/brain/awt320. Epub 2013 Nov 25. PMID 24277718
- [Result] Sances G, Tassorelli C, Pucci E, Ghiotto N, Sandrini G, Nappi G. Reliability of the nitroglycerin provocative test in the diagnosis of neurovascular headaches. Cephalalgia. 2004 Feb;24(2):110-9. doi: 10.1111/j.1468-2982.2004.00639.x. PMID 14728706
- [Result] Tassorelli C, Joseph SA, Buzzi MG, Nappi G. The effects on the central nervous system of nitroglycerin--putative mechanisms and mediators. Prog Neurobiol. 1999 Apr;57(6):607-24. doi: 10.1016/s0301-0082(98)00071-9. PMID 10221784